CLINICAL TRIAL: NCT01950949
Title: The Correlational Study of Pulse Pressure Variation in Various Tidal Volume in Mechanically Ventilated Patients Under General Anaesthesia
Brief Title: The Correlational Study of PPV in Various VT in Mechanically Ventilated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yi Liu (Other)
Responsible Party: Sponsor-Investigator, Yi Liu, Attending of AOC, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: plaghaoc001
Record Dates: First submitted 2013-07-26; First posted 2013-09-26 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Respiration, Artificial
MeSH Terms: conditions — Respiratory Aspiration | interventions — Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- change respiratory parameters, volume expanding (Experimental)
  Interventions: Other: 300 ml Hydroxyethyl Starch 130/0.4 and Sodium Chloride Injection infusing in 15 minutes if PPV under VT 8 ml/kg was larger than 13% in the initial investigation

INTERVENTIONS:
Other: 300 ml Hydroxyethyl Starch 130/0.4 and Sodium Chloride Injection infusing in 15 minutes if PPV under VT 8 ml/kg was larger than 13% in the initial investigation

SUMMARY:
Mesquida, J et al showed there was a significant linear correlation between pulse pressure variations under tidal volume 6 ml/kg and 8 ml/kg in patients after the resuscitation phase of severe sepsis and septic shock. No study revealed the actual relationship between various PPV under different VT. So we hypothesized that there were relationship between various PPV in different tidal volume settings. The objective of this study was to examine the relationship between various PPV.

ELIGIBILITY:
Inclusion Criteria:

scheduled for elective abdominal surgeries ASA (American Society of Anesthesiologists) I or II BMI 18-25 preoperative examination is normal

Exclusion Criteria:

acute lung injure acute respiratory distress syndrome cardiovascular diseases neurological disease renal or hepatic disease diabetes mellitus BMI less than 18 kg/m2 or greater than 25 kg/m2

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2012-07; Primary Completion 2014-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
invasive arterial blood pressure as a Measure of Safety | Day 1
  if instability of circulation, stop the clinical trial

REFERENCES:
- [Derived] Liu Y, Lou JS, Mi WD, Yuan WX, Fu Q, Wang M, Qu J. Pulse pressure variation shows a direct linear correlation with tidal volume in anesthetized healthy patients. BMC Anesthesiol. 2016 Sep 8;16:75. doi: 10.1186/s12871-016-0233-y. PMID 27609188